CLINICAL TRIAL: NCT02025465
Title: Randomized Trial Comparing Diltiazem and Metoprolol For Atrial Fibrillation Rate Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, William Carter, Professor of Medicine - West Virginia University, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1997386
Record Dates: First submitted 2013-12-16; First posted 2014-01-01 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Atrial Flutter; Metoprolol; Diltiazem
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Metoprolol; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoprolol (Experimental): Metoprolol 2.5 to 5.0 mg IV bolus over two minutes
  Repeat every five minutes up to a total dose of 15 mg as long as tolerated (Blood pressure is over 100 mm /Hg systolic (or BP is 90 to 100 mm\Hg systolic and the patient is not dizzy))
  If rate inadequate the physician has option of:
  1. Further doses of metoprolol IV or PO
  2. Intravenous amiodarone
  3. IV diltiazem
  4. Observation
  Interventions: Drug: Metoprolol
- Diltiazem (Active Comparator): Bolus 0.25 Mg/Kg over two minutes (average adult dose 20 mg).
  If after 15 minutes
  1. The first dose is tolerated, and
  2. Ventricular rate is over 100 beats a minute AND
  3. Blood pressure is over 100 mm /Hg systolic (or BP is 90 to 100 mm\Hg systolic and the patient is not dizzy)
  Give diltiazem 0.35 Mg/Kg over two minutes (average adult dose 25 mg).
  After initial bolus', start infusion 5 to 15 Mg/hour to maintain rate control as long as:
  1. BP over 100 mm/Hg or between 90 and 100 mm/Hg and the patient is not dizzy.
  If rate inadequate the physician has an option of:
  1. Metoprolol PO (by mouth) or IV (intravenous)
  2. Digoxin PO or IV
  3. Intravenous amiodarone
  4. Observation
  Interventions: Drug: Diltiazem

INTERVENTIONS:
Drug: Metoprolol — The attending ED physician may use higher or lower intravenous doses depending on patient response as this is the norm in clinical practice for these two medications used for decades for AF/FL rate control.
  Conversion of intravenous to oral, chronic management will be left to the discretion of the ED or managing medical team.
  Other Names: Lopressor
  Arms: Metoprolol
Drug: Diltiazem — The attending ED physician may use higher or lower intravenous doses depending on patient response as this is the norm in clinical practice for these two medications used for decades for AF rate control.
  Conversion of intravenous to oral medication for rate control for chronic management will be left to the discretion of the ED or managing medical team.
  Other Names: Cardizem
  Arms: Diltiazem

SUMMARY:
Atrial Fibrillation and atrial flutter (AF/FL) is the usually irregular beating of the heart and is a rapidly growing cause of hospitalization. Between 1993 to 2007 AF/FL hospitalizations have increased 203% compared to a 71% increase for all hospitalizations. Changing procedure management such as ablation, transesophageal have had a minimal impact on the trends and there is a need to evaluate Emergency Department (ED) management options of AF/FL that may decrease hospitalizations.

The most commonly used medications to control heart rate are metoprolol (MET), a beta blocker, or diltiazem (DT), a calcium channel blocker. Beta blockers are medications that cause the heart to beat more slowly and with less force. DT also helps blood vessels open up to improve blood flow. Both DT and MET are used alone or together with other medicines to treat severe chest pain (angina), high blood pressure (hypertension) or rapid heartbeat. Both are equally acceptable according to recent guidelines for AF/FL. There are limited studies comparing MET to DT for rate control for AF/FL.

The initial goal for AF/FL management in the Emergency Department is usually rate control.

The most commonly used rate control medications are metoprolol (MET), a beta blocker, or diltiazem (DT) a calcium blocker. Three major guidelines, including the American College of Cardiology (ACC) and the American Heart Association (AHA) indicate beta blockers and DT are equally acceptable medications for rate control in AF (3,4,5) assuming no contraindications.

There are limited studies comparing beta blockers (BB) to DT for rate control for AF:

1. Demircan, et. al., compared bolus intravenous BB and DT in 40 patients over a 20 minute period. No follow-up information after 20 minutes was reported. No attempt was made to look at intermediate or long term results. No patients converted to normal sinus rhythm over this short treatment period and there was slightly more rate decrease at 20 minutes, with DT versus BB (6).
2. Time from medication administration to heart rate and rhythm control. Additionally, currently guidelines consider BB or DT medications to slow AF/FL; however, there are some suggestions that BB may not only slow heart rate in AF/FL (as does DT) but also increase all AF/FL conversion from AF/FL to normal sinus rhythm(2), and aid in maintaining normal sinus rhythm (NSR) after cardioversion (10). With recent onset AF/FL occurring within 48 hours prior to the arrival to the ED, approximately 50% of AF/FL patients convert to normal rhythm spontaneously within 24 hours after arrival to the ED (6), making evaluation of current limited studies difficult. Thus, the investigators wish to examine the effect of initial medication strategy on time to NSR in a larger sample than has been previously performed.
3. A randomized study of 48 patients in China reported significantly slower heart rate up to 20 minutes with DT 10mg IV versus metoprolol 5mg IV but not after 30 minutes (7).
4. A retrospective study of post-operative coronary bypass patients showed the intravenous administration of the BB, esmolol, to be more effective than DT for rate control and conversion of AF/FL (8).
5. Hassan et al reported no difference in conversion to regular rhythm with esmolol verses DT in a small, under powered, randomized study of fifty ED patients (9). Conversion to sinus rhythm occurred in 10 patients (42%) in the DT group compared with 10 patients (39%) in the esmolol group (P = 1.0). There were no statistically significant differences in heart rate between the two medications at 1, 6, 12, and 24 hours after initiation of esmolol or DT infusion.

Examples of such well quoted strategy trials are the COURAGE trial published in the New England Journal of Medicine and the PROMISE Trial, a worldwide multi-centered study that is nearing completion goal of 10,000 patients of which, Charleston Area Medical Center (CAMC) has enrolled approximately 100 patients. In this trial, patients being evaluated for chest pain will be randomized to two treatment strategies and subsequent outcomes will be recorded.

Strategy trials do not attempt to manage treatment after an initial management strategy has been determined by randomization, but, whether the initial treatment affects long-term outcomes.

This will be a prospective, randomized study comparing the outcomes of a strategy using either MET or DT in patients with AF presenting to the Charleston Area Medical Center (CAMC) ED. After presentation and receiving consent, the patient will be randomized to receive either MET or DT.

DETAILED DESCRIPTION:
If either an initial DT or MET strategy are shown to be more effective in obtaining rate and rhythm control, decreasing length of stay in the ED, and decreasing admissions and readmissions, there is a potential for: 1.) Major health cost savings; 2.) Improved bed utilization for our hospital, which is frequently at capacity and unable to accept transfers from outlying hospitals; and, 3.) Education of ED and non-ED health care providers of optimal AF/FL medication options.

Sample

Preliminary information obtained from CAMC's Data Warehouse from July 1, 2011 to June 30, 2012 revealed 370 patients were seen in the Emergency Department (ED) at either CAMC Memorial or General Hospitals with a diagnosis of AF/FL, without any other acute co-morbidity. The investigators will identify which Hospital the patient was enrolled.

The investigators will enroll a total of 150 patients based on the following:

Prior data indicate that the conversion to a normal sinus rhythm by 8 hours is approximately 20%. If the investigators wish to detect a 25% change between medications then the investigators would need to include a total of 150 patients (75 in each cohort) to reject the null hypothesis that the conversion rates are equal between the 2 medications with probability (power) 0.8 and Type I error < 0.05. The investigators will use a continuity-corrected chi-squared statistic or Fisher's exact test to test our hypothesis. Power analysis performed using GPower Version 3.

Procedures

Potential study patients will be identified by an ED nurse or a member of the study team using the inclusion and exclusion criteria. ED nurses will be informed of the study by charge nurses who have been educated about the protocol by the research team. The purpose, content and logistics of the study will also be described to ED physicians participating in the study. Research assistants, when available, will be notified by cell phone or pager to see patient in the ED within 20 minutes. The attending physician or resident will be informed of the potential study patient. The attending physician or resident will give the research associate/member of the study team permission to discuss the study with the patient. If the patient is interested in participating in the study, the research associate/member of the study team will discuss the details of the study and review the consent form. It is likely the onset of treatment with DT or MET will be delayed 30 to 40 minutes due to the consenting process and study enrollment. The attending physician must agree to this delay.

At this point the attending physician will discuss the study with the patient and answer questions. The physicians or resident initially talking with the patients about being in the trial will have Collaborative Institutional Training Initiative (CITI) training. General education to the ED staff will be made concerning aims and objectives of the strategy study. If the patient is still interested and willing to participate, the informed consent and Health Insurance Portability and Accountability Act (HIPAA) privacy statement will be signed.

Following consent, patients will be randomized to either IV diltiazem (DT) or IV metoprolol (MET). Sealed envelopes containing the randomized treatment protocol will be maintained on the ED premises to be pulled consecutively after a patient has been consented to be in the study. Inside the envelope, the specific treatment plan will be revealed. Treatment with either DT or MET will be initiated using standard CAMC protocol. Deviations from the randomly assigned medication regimen would be at the attending physician's discretion pending vital signs response. If the study drug is stopped or changed to a different type of medication, the patient's participation will continue and medications will be documented with the analysis of results being the intent to treat.

The same physicians rotate at both General and Memorial Hospitals. The investigators will start at the Memorial Hospital, but after experience with enrollment the investigators may enroll patients from both Hospitals.

Data Analysis

Basic descriptive statistics including means and standard deviations for continuous variables and proportions and frequencies for categorical variables will be used to describe the patient sample and disease characteristics.

To determine if a medication regimen (MET vs DT) is noted by descriptive analysis to be associated with primary aim 1 for treating AF/FL in the ED or during hospitalization (Primary Aim-1), the investigators will describe the proportion of patients with rhythm control (defined as normal sinus rhythm) by time of ED discharge using Chi-square analysis with continuity correction. Using the same statistical tests, the investigators will describe the proportion of patients with normal sinus rhythm at time of hospital discharge, in patients admitted to CAMC. Possible confounders, including patient characteristics, co-morbid conditions, ED events, or deviation from medicine regimen on achieving NSR will be examined by comparing patients with the confounder to those without the confounder of interest using Chi-square with continuity correction analyses if data is categorical, t-test or Mann-Whitney U analysis if data is continuous. In addition, the investigators will examine the effect of medication regimen on rate control (defined as heart rate < 100 bpm) (Primary Aim-2) at 2, 4, 6, 8 hours in the identical manner as described for rhythm control including the examination of confounding variables.

The proportion of patients receiving CAMC hospital admission versus discharged to home from the ED will be described between the two medication regimens using Chi-square analysis with continuity correction to determine if one regimen resulted in a greater percentage of home discharges directly from the ED (Secondary Aim-1). The effect of possible confounders including patient characteristics, ED events, achieving rate and/or rhythm control in the ED or deviation from medication regimen will be examined by describing patients with the confounder to those without the confounder of interest on the need for hospital admission using Chi-square with continuity correction analyses if data is categorical, t-test or Mann-Whitney U analysis, if data is continuous. Those confounders that are shown to associate with ED discharge to home will be included in a multivariate analysis (binomial logistic regression) to examine if medication regimen associates with ED discharge to home in the presence of confounders.

To determine if a medication regimen (MET vs DT) associated with decreased financial costs (Secondary Aim-2), ED costs will be examined between the 2 medication regimens in all patients using t-tests, or Mann-Whitney U analysis. In addition, the total cost of hospitalization (ED + hospital costs) of patients admitted to the CAMC hospital from the ED will be examined between the medication regimens. Cost will also be examined in relationship to length of stay by examining cost /length of stay between the two treatment groups using the same statistical tests.

The need for readmission and atrial fibrillation reoccurrence as reported by the phone questionnaire (Secondary Aim-3) will be compared between the two medication regimens using Chi-square with continuity correction analyses. The investigators will also determine which rate control medication at time of phone interview associates with freedom from atrial fibrillation reoccurrence using chi-square analysis. Lastly, the time between discharge and phone survey study completion (maximum: 6 months) will be determined and the investigators will examine the effect of this lag time (4- 6 months) on the percentage of patients requiring readmission and/or having a reoccurrence of atrial fibrillation via chi square analysis.

For all applicable analyses described above, Fisher's exact tests will be substituted for Chi square analysis when appropriate. For all comparisons, a p level of < 0.05 will be used to determine statistical significance. The statistical package Statistical Analysis Software (SAS) (Version 9.3) will be used to analyze data.

Confidentiality

Minimal patient identification information will be collected. The patient account number and telephone number must be collected. Subjects will also be assigned a study number for data analysis; account numbers will not be included in the data analysis. Personal health information will be available only to the study investigators. All collected data will be stored in a locked filing cabinet in the Emergency Department until it can be delivered to CAMC Outcomes Research. Electronic data will be stored on a password protected computer. At the conclusion of the study, all data collection sheets will be shredded and electronic data destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Charleston Area Medical Center (CAMC) General or Memorial Hospital ED with a primary diagnosis of AF/FL
* Patients with a mean ventricular rate of 100 beats per minute or more within one hour of presentation

Exclusion Criteria:

* Under age 18 years
* A diagnosis of acute coronary syndrome (ACS) made by the admitting ED physician (ST elevation myocardial infarction, non-ST elevation myocardial infarction, unstable angina) (beta blockers are a Class I medications for ACS)
* Known history of heart failure with an ejection fraction <50%
* Known ejection fraction <45%, regardless of a history of heart failure. Heart failure and a history of heart failure with an ejection fraction of 40-50% may occur with a normal ejection fraction now referred to as Heart Failure With Preserved Ejection Fraction (HFpEF) or "diastolic dysfunction". A low ejection fraction is not always associated with heart failure. Our technology of measuring ejection fraction is by no means perfect. It is acceptable to use MET in larger than usual starting doses of MET for rate control or patients with "diastolic dysfunction", but not systolic dysfunction. Thus, a patient who has an ejection fraction of 42% may possibly have an ejection fraction of 37%, possible lower. Thus the investigators want to avoid the possibility of a patient with a history of heart failure does not receive MET unless the investigators feel systolic heart failure is not present.
* Systolic blood pressure <90 mm Hg or between 90-99 AND patient is experiencing symptoms of dizziness
* Known allergy or adverse reactions to diltiazem or metoprolol. This is very rare.

Exclusions from ECG readings:

* Current Atrioventricular (AV) block (2nd or 3rd degree)
* Pre-excitation syndromes - Wolfe Parkinson White (WPW) (Accelerated AV conduction- a rare condition where MET and DT are not advised)
* Pulse rate less 100/minute on ED admission (already at rate control)
* Cardiogenic shock or heart failure requiring inotropic agents or intubation
* Respiratory failure requiring intubation
* Pregnancy or lactation (neither pregnancy or lactation are listed as definitely safe for either medication)
* Asthma, defined as (asthma is a relative contraindication for MET:
* current use of inhaler
* use of steroids for dyspnea
* history of being treated for asthma
* Inability or unwillingness to provide informed consent
* Physician decision
* If either medication is a relative contraindication, the patient cannot be randomized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Conversion to sinus rhythm | 2 hours
  Conversion to sinus rhythm
Conversion to sinus rhythm | 4 hours
  Conversion to sinus rhythm
Conversion to sinus rhythm | 6 hours
  Conversion to sinus rhythm
Conversion to sinus rhythm | 8 hours
  Conversion to sinus rhythm
Heart rate control | 2 hours
  Heart rate control
Heart rate control | 4 hours
  Heart rate control
Heart rate control | 6 hours
  Heart rate control
Heart rate control | 8 hours
  Heart rate control

SECONDARY OUTCOMES:
Home discharges from Emergency Department (ED) | Date of admission to ED and duration of hospital stay, an expected average of 5 weeks.
  Home discharges from Emergency Department (ED)
Total hospital cost | Date of admission to ED and duration of hospital stay, an expected average of 5 weeks.
  Total costs during the time in the ED plus any in hospital costs that might have occurred.
Rehospitalization for Atrial Fibrillation | Up to 6 months post discharge
  Rehospitalization for Atrial Fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: William H. Carter, MD, Principal Investigator — West Virginia University - Charleston Division/CAMC; Bill Payne, MD, Study Director — West Virginia University - Charleston Division/CAMC
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong CX, Brooks AG, Leong DP, Roberts-Thomson KC, Sanders P. The increasing burden of atrial fibrillation compared with heart failure and myocardial infarction: a 15-year study of all hospitalizations in Australia. Arch Intern Med. 2012 May 14;172(9):739-41. doi: 10.1001/archinternmed.2012.878. No abstract available. PMID 22782205
- [Background] Wolowacz SE, Samuel M, Brennan VK, Jasso-Mosqueda JG, Van Gelder IC. The cost of illness of atrial fibrillation: a systematic review of the recent literature. Europace. 2011 Oct;13(10):1375-85. doi: 10.1093/europace/eur194. Epub 2011 Jul 14. PMID 21757483
- [Background] Stiell IG, Macle L; CCS Atrial Fibrillation Guidelines Committee. Canadian Cardiovascular Society atrial fibrillation guidelines 2010: management of recent-onset atrial fibrillation and flutter in the emergency department. Can J Cardiol. 2011 Jan-Feb;27(1):38-46. doi: 10.1016/j.cjca.2010.11.014. PMID 21329861
- [Background] Lip GY, Huber K, Andreotti F, Arnesen H, Airaksinen JK, Cuisset T, Kirchhof P, Marin F; Consensus Document of European Society of Cardiology Working Group on Thrombosis. Antithrombotic management of atrial fibrillation patients presenting with acute coronary syndrome and/or undergoing coronary stenting: executive summary--a Consensus Document of the European Society of Cardiology Working Group on Thrombosis, endorsed by the European Heart Rhythm Association (EHRA) and the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2010 Jun;31(11):1311-8. doi: 10.1093/eurheartj/ehq117. Epub 2010 May 6. PMID 20447945
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Kay GN, Le Huezey JY, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann LS, Smith SC Jr, Priori SG, Estes NA 3rd, Ezekowitz MD, Jackman WM, January CT, Lowe JE, Page RL, Slotwiner DJ, Stevenson WG, Tracy CM, Jacobs AK, Anderson JL, Albert N, Buller CE, Creager MA, Ettinger SM, Guyton RA, Halperin JL, Hochman JS, Kushner FG, Ohman EM, Stevenson WG, Tarkington LG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force. 2011 ACCF/AHA/HRS focused updates incorporated into the ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2011 Mar 15;123(10):e269-367. doi: 10.1161/CIR.0b013e318214876d. Epub 2011 Mar 7. No abstract available. PMID 21382897
- [Background] Demircan C, Cikriklar HI, Engindeniz Z, Cebicci H, Atar N, Guler V, Unlu EO, Ozdemir B. Comparison of the effectiveness of intravenous diltiazem and metoprolol in the management of rapid ventricular rate in atrial fibrillation. Emerg Med J. 2005 Jun;22(6):411-4. doi: 10.1136/emj.2003.012047. PMID 15911947
- [Background] Diao, Hong-ying; Liu, Bin; Chen, Hong-Bo; Shi, Yong-feng; Wang, Li-juan. Comparison of the effectiveness of intravenous diltiazem and metoprolol in controlling the rapid ventricular rate in patients with atrial fibrillation. Journal of Emergency Medicine 2009; Vol. 18: 1085-87
- [Background] Hilleman DE, Reyes AP, Mooss AN, Packard KA. Esmolol versus diltiazem in atrial fibrillation following coronary artery bypass graft surgery. Curr Med Res Opin. 2003;19(5):376-82. doi: 10.1185/030079903125001929. PMID 13678474
- [Background] Hassan S, Slim AM, Kamalakannan D, Khoury R, Kakish E, Maria V, Ahmed S, Pires LA, Kronick SL, Oral H, Morady F. Conversion of atrial fibrillation to sinus rhythm during treatment with intravenous esmolol or diltiazem: a prospective, randomized comparison. J Cardiovasc Pharmacol Ther. 2007 Sep;12(3):227-31. doi: 10.1177/1074248407303792. PMID 17875950
- [Background] Kuhlkamp V, Schirdewan A, Stangl K, Homberg M, Ploch M, Beck OA. Use of metoprolol CR/XL to maintain sinus rhythm after conversion from persistent atrial fibrillation: a randomized, double-blind, placebo-controlled study. J Am Coll Cardiol. 2000 Jul;36(1):139-46. doi: 10.1016/s0735-1097(00)00693-8. PMID 10898425